CLINICAL TRIAL: NCT00074451
Title: Genomewide Search for Loci Underlying Metabolic Syndrome
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1241; R01HL073882 (NIH)
Record Dates: First submitted 2003-12-12; First posted 2003-12-15 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2008-08

CONDITIONS: Metabolic Syndrome X; Cardiovascular Diseases; Heart Diseases; Obesity; Hypertension; Hyperinsulinism; Insulin Resistance
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases; Heart Diseases; Obesity; Hypertension; Hyperinsulinism; Insulin Resistance

SUMMARY:
To identify the genes involved in the metabolic syndrome.

DETAILED DESCRIPTION:
BACKGROUND:

Metabolic syndrome, characterized by clustering of multiple metabolic abnormalities including abdominal obesity, dyslipidemia, hyperinsulinemia, hyperglycemia, and hypertension, is one of the most important risk factors for cardiovascular disease and stroke. Genetics play a significant role in determining the individual susceptibility to metabolic syndrome and the inter-individual variation in its associated phenotypes, though these genetic factors remain largely unknown. The long-term goal is to identify the metabolic syndrome susceptibility genes and their functional variants.

DESIGN NARRATIVE:

The goal of the research is to study the underlying phenotypic structure of the metabolic syndrome and to systematically search for genetic loci predisposing to the metabolic syndrome using the genome scan approach. The specific aims are: (1) to screen about 10,000 sibling pairs aged 40 to 64 years in Anqing, Anhui China, on intermediate phenotypes of the metabolic syndrome including body mass index, waist and hip circumference, serum lipid profiles (triglyceride, HDL-, LDL-, and total cholesterol), fasting serum glucose and insulin level, and blood pressure; (2) to study the underlying phenotypic structure of the metabolic syndrome in the about 10,000 ascertained sibling pairs using factor analysis; (3) to select and genome scan 800 nuclear families from the pool of the ascertained sibling pairs using Weber screening set 10 markers. Each selected nuclear family contains a "proband" and >=3 other family members. The values of the three most significant factors for metabolic syndrome in the factor analysis (see specific aim 2) will be used to classify "proband" status for each subject. A "proband" is defined as having >=2 out of 3 factor values falling into the same side of the 10/90 percentile tails of the corresponding age- and sex-adjusted population distributions; (4) to test for linkage in the genome-scanned families on intermediate phenotypes and factors of metabolic syndrome using the Unified Haseman-Elston method. In addition to the univariate test, linkage analysis will be performed using a novel multivariate version of the Unified H-E method, which has recently been proposed and shown to be significantly more powerful than the univariate test for traits with common genetic determinants; (5) to perform expansion or replication linkage studies on loci identified in the genome scan in 300-400 additional families with >=1 proband with a denser set of markers.

ELIGIBILITY:
No eligibility criteria

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2003-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xu Xin, Principal Investigator — Harvard School of Public Health (HSPH)